CLINICAL TRIAL: NCT00843310
Title: Phase II Study of Revlimid (Lenalidomide), Melphalan, and Dexamethasone (ReMeDex) for Newly Diagnosed Multiple Myeloma Patients Not Undergoing Autologous Transplantation
Brief Title: Combination of Revlimid, Melphalan and Dexamethasone as First Line Treatment for Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: NYU Langone Health (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-919; Celgene # RV-MM-PI-289 (Other: Celgene)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; frontline treatment; first-line treatment
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Melphalan; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ReMeDex (Experimental): Treatment phase (28 days/cycle x 6 cycles):
  Lenalidomide: 10 mg/day orally on days 1-21, followed by 7 days of rest. Melphalan: 4 mg/m2 daily on days 1-4. Dexamethasone: 40 mg daily on days 1, 8, 15 and 22.
  Maintenance Phase (for subjects who achieve partial response or better at the end of the treatment phase):
  lenalidomide: 10 mg/day orally on days 1-21 followed by 7 days of rest (28 days/cycle) for a maximum of 24 cycles.
  Interventions: Drug: Lenalidomide (Revlimid); Drug: Melphalan; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide (Revlimid)
  Other Names: Revlimid
Drug: Melphalan
Drug: Dexamethasone

SUMMARY:
This study is to determine whether addition of Revlimid to standard therapy will increase overall and complete response rates compared to historical standard frontline therapy and whether this combination treatment has fewer side effects than similar combination induction treatment.

DETAILED DESCRIPTION:
Current multiple myeloma therapies, typically an induction regimen followed by consolidation therapy with high dose chemotherapy and autologous stem cell rescue (autologous transplantation), can induce remission but relapse and death are inevitable. A growing body of literature suggests that consolidation therapy with autologous transplantation does not confer additional survival benefit and may have increased procedure-related morbidity and mortality in patients over 65 years old. Autologous transplantation is no longer recommended as standard care for this population. In addition, certain patients may not be eligible for autologous transplantation due to co-morbid medical conditions or may elect not to undergo the procedure for personal reasons.

The historic standard of care for multiple myeloma patients who were not eligible for autologous transplantation for consolidation was induction therapy with melphalan/ prednisone (MP), often followed by some form of maintenance therapy after achievement of complete or partial remission. A recent phase 3 study showed that the addition of thalidomide to MP (MPT) demonstrated higher overall and complete response rates. For patients who are eligible for autologous transplantation, thalidomide/ dexamethasone (Thal Dex) induction therapy is considered the standard of care, but a phase 2 study of lenalidomide (Revlimid)/ dexamethasone (Rev Dex) induction therapy demonstrated higher overall and complete response rates compared to Thal Dex. In addition, lenalidomide has a favorable side effect profile compared to thalidomide. Based on these data, we hypothesize that the combination of Revlimid/ melphalan/ dexamethasone (ReMeDex) induction therapy for myeloma patients who are not planned for autologous transplantation due to age restriction or other factors may demonstrate higher overall and/ or complete response rates with fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Newly Diagnosed multiple myeloma, ISS stage I-III requiring therapy: Serum M-protein ≥1 gm/dL (≥10 gm/L), Urine M-protein ≥200 mg/24 hr, Serum FLC assay: involved FLC ≥10 mg/dL (≥100 mg/L) provided serum FLC ratio is abnormal
* Previously untreated except prior treatment with corticosteroid less than one full cycle of pulsed dose dexamethasone (40 mg daily days 1-4, 9-12, and 17-20) or equivalent is allowed. Concomitant administration of IV bisphosphonates, Zometa (zoledronic acid, up to 4 mg IVSS over 30 minutes every four weeks) or Aredia (alendronate, up to 90 mg IVSS over 4 hours every four weeks), for prophylaxis against skeletal complications due to lytic bone disease or for acute management of hypercalcemia is allowed. Concomitant external beam radiation therapy for local management of lytic bone disease is allowed.
* Age ≥ 18 years old
* Life expectancy ≥ 12 weeks
* Eastern Cooperative Oncology Group (ECOG) Performance Status will be employed. ECOG 0-2 accepted.
* WBC ≥ 3.0 X 103/ µL, ANC ≥ 1.5 X 103/ µl, Hgb ≥ 8.0 gm/ dL, Plt ≥ 75 X 103/ µl, Serum Creatinine ≤ 2.0 mg/ dL
* Ability to understand and the willingness to sign a written informed consent document.
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix A: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

* Prior therapy with Revlimid®, Thalomid (thalidomide), Velcade (bortezomib), Alkeran (melphalan) excluded. Prior therapy with corticosteroid allowed as defined in inclusion criteria.
* No prior or concurrent treatment with an investigational agent.
* Active Hepatitis B or C excluded, New York Heart Association grade III/IV congestive heart failure excluded, History of bleeding disorder excluded, History of platelet function disorder, History of deep vein thrombosis or other thromboembolic event excluded
* Prior history of allergic reaction to IMiD™ compounds (Thalidomide, Lenalidomide) excluded.
* Concomitant treatment with nonsteroidal antiinflammatory drugs (NSAIDs)(with the exception of aspirin) or other nephrotoxic agents is excluded.
* Serum creatinine > 2.0 mg/ dL is excluded
* Pregnancy and breastfeeding excluded
* Known HIV+ patients are excluded.
* Other active hematologic or solid tumor or history of such disease requiring therapy of any form within five years of screening is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hearn J Cho, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Bellevue Hospital, New York, New York
  - NYU Cancer Center, New York, New York
  - NYU Tisch Hospital, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from NYU medical center and its affiliated hospitals from Dec 2008 through Apr 2011.
Pre-assignment Details: Total 8 patients were enrolled. One patient withdrew before the treatment started.
Period: Overall Study
Arm/Group | ReMeDex
Started | 8
Completed | 1
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | ReMeDex
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 69 [67 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race/Ethnicity, Customized [Number; unit: paticipants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Toxicity, Time to Progression & Progression Free Survival
Description: Toxicity will be scored using CTCAE version 3.0 for toxicity and adverse event reporting.
  Progressive Disease: requires any one or more of the following:
  1. Increase of ≥25% from baseline in Serum M-component and/or (the absolute increase must be ≥0.5 g/dl)b
  2. Urine M-component and/or (the absolute increase must be ≥200 mg/24 h
  3. Only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels. The absolute increase must be >10 mg/dl.
  4. Bone marrow plasma cell percentage: the absolute % must be ≥10%c
  5. Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
  6. Development of hypercalcemia (corrected serum calcium >11.5 mg/dl or 2.65 mmol/l) that can be attributed solely to the plasma cell proliferative disorder
Time Frame: every 28 days during therapy and every month after therapy for 2 years
Population: No data are available because data were not collected. Pi left the institution and slow accrual did not allow for sufficient data collection prior to PI leaving institution. No data were analyzed.
Arm/Group | ReMeDex
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Only 7 out of 8 patients were treated. The percentage of affected patients was based on those 7.
Arm/Group | ReMeDex
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReMeDex (N=7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pain-back (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReMeDex (N=7)
Abdominal pain or cramping (Gastrointestinal disorders) | 1
Alkaline phosphatase (Investigations) | 1
Anorexia (Gastrointestinal disorders) | 3
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Constitutional Symptoms-Other (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 1
Diarrhea patients without colostomy (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Edema (Vascular disorders) | 1
Fatigue (lethargy, malaise, asthenia) (General disorders) | 3
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 1
Gastrointestinal-Other (Gastrointestinal disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Infection without neutropenia (Infections and infestations) | 1
Musculoskeletal-Other (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Pain-Other (General disorders) | 2
Platelets (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Thrombosis/embolism (Vascular disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes